CLINICAL TRIAL: NCT06017908
Title: Identification of Visual Dependence in PPPD Patients With an Enhanced Rod and Disc Test (RDT) and Optokinetic After Nystagmus (OKAN) With the Aid of Virtual Reality.
Brief Title: Identification of Visual Dependence in PPPD Patients With the Aid of Virtual Reality.
Acronym: OKAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23079_OKAN
Record Dates: First submitted 2023-03-15; First posted 2023-08-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-03

CONDITIONS: PPPD
Keywords: Virtual Reality; PPPD; Rod and Disc Test; Optokinetic after nystagmus; Visual dependence

STUDY DESIGN:
Intervention Model Description: Intervention of the Virtual Reality goggles will be evaluated in a small clinical trial to determine the feasibility of the product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPPD patients (Experimental): Virtual Reality will be used to execute the RDT and OKAN in PPPD patients.
  Interventions: Device: Optokinetic stimulation through Virtual Reality
- Healthy patients (Experimental): Virtual Reality will be used to execute the RDT and OKAN in healthy PPPD patients.
  Interventions: Device: Optokinetic stimulation through Virtual Reality

INTERVENTIONS:
Device: Optokinetic stimulation through Virtual Reality — The experiment will be conducted in two phases. In the first experiment the patients will be passively watch the visual images while seated. An optokinetic stimulus will be delivered through the VR headset by displaying rotating visual patterns. In the second trial they will have to perform the enhanced rod and disc test.

SUMMARY:
The aim of this study is to evaluate whether increased visual dependence can be identified with the help of Virtual Reality (VR). Increased visual dependence is a general term for patients with increased dependence on vision in maintaining their balance. Patients suffering from persistent postural perceptual vertigo (PPPD) often suffer from increased visual dependence. This in turn leads to complaints such as visual vertigo, agoraphobia and fear of falling. Visual dependence is normally measured using the optokinetic after nystagmus (OKAN) and the rod and disc test (RDT). In this study, these two tests are performed with the aid of Virtual Reality.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether increased visual dependence can be identified with the help of Virtual Reality (VR). Visual dependence is normally measured using the optokinetic after nystagmus (OKAN) and the rod and disc test (RDT). In this study, these two tests are performed with the aid of Virtual Reality. The OKAN is measured by eye tracking, a key item already used daily in instruments such as video nystagmography (VNG) and video head impulse test (vHIT). Another test representative of visual dependence is the Rod and Disc test (RDT). In the RDT, patients are asked to complete a visual task so that researchers gain more knowledge about visual dependence. Until now, these tests have been performed using a large set-up and many different materials. Moreover, the exact underlying mechanism of visual dependence in PPPD patients is still unknown. The aim of this study is to investigate whether Virtual Reality can be a useful tool when performing the OKAN and RDT. In this way, a better understanding of visual dependence is sought. This study aims to determine the normative values for the OKAN and RDT performed with the aid of Virtual Reality. Therefore, a healthy group of individuals will be compared with PPPD patients as they suffer from visual dependence. To evaluate the effectiveness of the OKAN and RDT via VR, the results will be compared with the scores of the visual vertigo analogue scale (VVAS), a questionnaire to assess visual dependence.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic vertigo (>3 months)

Exclusion Criteria:

* Minors
* Patients with a history of epilepsy.
* Patients with an alcohol use disorder

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Device feasibility | 1 year
  Time constant and velocity of eye movements

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Topsakal, Prof, MD, Principal Investigator — Free University of Brussels
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No